CLINICAL TRIAL: NCT02988388
Title: Lung Tissue Research Consortium
Acronym: LTRC
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: LTR01
Record Dates: First submitted 2016-12-07; First posted 2016-12-09 (Estimated); Last update posted 2019-03-08 (Actual); Status verified 2017-08

CONDITIONS: Chronic Obstructive Pulmonary Disease; Interstitial Lung Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — For a subset of LTRC participants who provide applicable consent, a portion of collected blood will be stored in a Paxgene DNA tube for DNA generation. DNA will be stored in a central laboratory and available for request by qualified researchers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lung biopsy/lobectomy: Adults ages 21 or older who are undergoing lung surgery for suspected malignancy or metastases.
  Interventions: Procedure: Lung biopsy/lobectomy

INTERVENTIONS:
Procedure: Lung biopsy/lobectomy — Lung biopsies and lobectomies are not experimental. Participants will undergo a lung biopsy or a lobectomy as part of standard of care.

SUMMARY:
The LTRC will facilitate histopathological research of pulmonary diseases by collecting lung tissues from donors and preparing and distributing collections of tissue specimens to researchers within and outside the LTRC. Collections of specimens will be linked to individual clinical data appropriate to the particular disease. The primary goal of the LTRC is to identify participants with suspected lung cancer or metastatic disease who are willing to provide informed consent for research use of their specimens and data. Secondarily, the LTRC investigators intend to collect clinical data, limited exposure data, physiologic studies, and radiographic studies from these participants.

ELIGIBILITY:
Inclusion Criteria:

* Adults ages 21 or older who are undergoing lung surgery for suspected malignancy or metastases.

Exclusion Criteria:

* Diagnosis of cystic fibrosis or pulmonary hypertension.
* Any other condition that, in the judgment of the investigator, precludes participation.
* Failure to obtain written consent.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults ages 21 or older who are undergoing lung surgery for suspected malignancy or metastases.
Sampling Method: Non-Probability Sample
Enrollment: 247 (Actual)
Dates: Start 2017-02-23 (Actual); Primary Completion 2019-01-28 (Actual); Study Completion 2019-02-21 (Actual)

PRIMARY OUTCOMES:
Clinical diagnosis | Two months following surgery
  A final diagnosis of the participant's lung disease will be rendered by the clinical center PI.

CONTACTS AND LOCATIONS:
Overall Officials: Tom Croxton, Study Director — National Heart, Lung, and Blood Institute (NHLBI)
Locations (4):
- United States (4):
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Temple University, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may submit an application for access to LTRC participant data including clinical and pathological diagnoses, radiological images (CT scans) and diagnoses, environmental and occupational exposure questionnaires, respiratory questionnaires and assessments, pulmonary function testing, concomitant therapy, medical history, smoking history, and laboratory measures. Gene array data are also available for a subset of participants. All data are de-identified. No protected health information is released to researchers external to LTRC.

REFERENCES:
- [Derived] Allen RJ, Stockwell A, Oldham JM, Guillen-Guio B, Schwartz DA, Maher TM, Flores C, Noth I, Yaspan BL, Jenkins RG, Wain LV; International IPF Genetics Consortium. Genome-wide association study across five cohorts identifies five novel loci associated with idiopathic pulmonary fibrosis. Thorax. 2022 Aug;77(8):829-833. doi: 10.1136/thoraxjnl-2021-218577. Epub 2022 Jun 10. PMID 35688625